CLINICAL TRIAL: NCT02582944
Title: Electromagnetic Navigation for Peripheral Pulmonary Lesions Using a Tip Tracked Steerable Catheter and Optical Guidance
Brief Title: Electromagnetic Navigation for Peripheral Pulmonary Lesions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201502080
Record Dates: First submitted 2015-10-20; First posted 2015-10-21 (Estimated); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: Peripheral Lung Lesions
MeSH Terms: interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Arm 1: Electromagnetic navigation (Experimental): * The bronchoscope will be inserted transorally into the tracheobronchial tree and a standard airway inspection will be performed.
  * Following airway inspection, the bronchoscope will be removed and the tip tracked steerable catheter with optical system will be advanced transorally through the vocal cords and into the tracheobronchial tree.
  * Once the tip tracked catheter has been advanced to the peripheral pulmonary target lesion, the optical SpinView system will be removed from the tip tracked catheter and the 1.4mm radial endobronchial ultrasound mini-probe will be inserted through the tip-tracked catheter into the lung periphery to confirm the presence of a peripheral pulmonary lesion and accurate navigation.
  * Once target confirmation has been performed using radial probe endobronchial ultrasound, biopsy of the peripheral lesion will be performed using biopsy forceps, brushes and aspiration needles.
  Interventions: Device: Olympus BF-180 bronchoscope (standard adult); Device: Veran Spinview Thoracic Navigation System; Device: Olympus UM-S20-17S; Procedure: Biopsy

INTERVENTIONS:
Device: Olympus BF-180 bronchoscope (standard adult) — -Standard of care
Device: Veran Spinview Thoracic Navigation System — -Electromagnetic navigation
Device: Olympus UM-S20-17S — -Endobronchial ultrasound mini-probe
Procedure: Biopsy

SUMMARY:
Despite technological advancements directed towards the diagnosis of peripheral pulmonary lesions, an optimal approach has yet to be designed. The potential advantages of catheter based techniques include the ability to utilize instruments smaller than the diameter of a conventional bronchoscope, thereby allowing better access to the lung periphery. The drawbacks of a catheter based approach include the relative inability to steer a conventional catheter, and the inability to perform direct visualization and airway inspection through a conventional catheter. This study will evaluate a novel steerable catheter system with optical capabilities and pair this with electromagnetic navigation bronchoscopy to biopsy peripheral pulmonary lesions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with peripheral lung lesions 1-7cm in size identified on chest CT with the intention to undergo bronchoscopic evaluation and biopsy. The decision to pursue biopsy will be made by the treating physician and agreed upon by the patient.
* Are at least 18 years old
* Are able to provide informed consent

Exclusion Criteria:

* Patients who refuse to participate
* Are less than 18 years of age
* Are pregnant
* Are physically unable to tolerate flexible bronchoscopy or moderate sedation as determined by the bronchoscopist
* Are unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-03-25 (Actual); Primary Completion 2017-05-19 (Actual); Study Completion 2017-05-19 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield of peripheral bronchoscopy using the tip tracked steerable catheter with removable optics and electromagnetic navigation guidance | At the time of procedure (1 day)
  -Primary outcome of diagnostic yield based on final cytology and/or histopathology will be determined from the results of the bronchoscopy. A biopsy that results in a specific diagnosis, either malignant or benign, that adequately explains the clinical scenario as determined by the treating physician, will be considered truly positive.

SECONDARY OUTCOMES:
Confirmation of successful navigation by using radial probe endobronchial ultrasound | At the time of procedure (1 day)
Safety as measured by adverse event rates | At the time of procedure (1 day)
  -Pneumothorax will be documented by post-biopsy CXR or chest ultrasonography, and the number requiring intervention, such as chest tube placement, will be recorded. Significant hemoptysis will be defined as bleeding noted at the time of procedure that requires a change in the level of care (e.g. outpatient to inpatient or inpatient to ICU) or a blood transfusion. Other adverse events that are common to bronchoscopy will be monitored

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Chen, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu